CLINICAL TRIAL: NCT04909619
Title: Suprazygomatic Maxillary Nerve Block in Cleft Palate Outcomes: Can we Minimize Analgesic and Opioid Use?
Brief Title: Suprazygomatic Maxillary Nerve Block in Cleft Palate Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-4219
Record Dates: First submitted 2021-03-12; First posted 2021-06-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cleft Palate Children
Keywords: Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided bilateral suprazygomatic maxillary nerve block (Experimental): Patients randomized to this arm will receive an ultrasound-guided bilateral suprazygomatic maxillary nerve block using 0.15 ml/kg of 0.2% ropivacaine per side, for a total of 0.3 ml/kg immediately after induction of general anesthesia and prior to incision. Participants will also receive local infiltration of the palate with an equivalent injection volume of 0.9% saline with 1:400,000 epinephrine at 2 ml/kg. Pediatric anesthesiologists with fellowship training in regional anesthesia will perform the nerve block. Local anesthetic infiltration will be performed by one of four board-certified pediatric plastic and craniofacial surgeons during repair of the palate. Patients, parents, surgeons, and the anesthesiologist will not be blinded to the specific intervention group due to the nature of the procedures involved. Nurses and the two key personnel responsible for data collection and analysis will be blinded throughout the entirety of the study.
  Interventions: Procedure: Ultrasound-guided bilateral suprazygomatic maxillary nerve block
- Local anesthetic infiltration of the palate (Active Comparator): Patients randomized to this arm will receive local infiltration of the palate using 0.125% bupivacaine + 1:400,000 epinephrine at a dose of 2 ml/kg intraoperatively. Local anesthetic infiltration will be performed by one of four board-certified pediatric plastic and craniofacial surgeons during repair of the palate. Patients, parents, surgeons, and the anesthesiologist will not be blinded to the specific intervention group due to the nature of the procedures involved. Nurses and the two key personnel responsible for data collection and analysis will be blinded throughout the entirety of the study.
  Interventions: Procedure: Local anesthetic infiltration of the palate

INTERVENTIONS:
Procedure: Ultrasound-guided bilateral suprazygomatic maxillary nerve block — The maxillary nerve, V2, is purely a sensory branch of the trigeminal nerve. V2 exits the skull through the foramen rotundum and courses through the pterygopalatine fossa, a small pyramid-shaped depression located posterior to the maxilla. As the maxillary nerve exits the pterygopalatine fossa, it divides into numerous branches that supply sensation to the posterior nasal cavity, palate, sinuses, and maxilla. It is within the pterygopalatine fossa that the maxillary nerve is targeted and anesthetized during the block. With the patient in the supine position after nasotracheal intubation, a needle is inserted perpendicularly between the upper border of the zygomatic arch and posterior orbital rim until it reaches the greater wing of the sphenoid, where the needle is then retracted by a few millimeters and redirected toward the nasolabial fold until it hits the pterygopalatine fossa.
  Arms: Ultrasound-guided bilateral suprazygomatic maxillary nerve block
Procedure: Local anesthetic infiltration of the palate — Local anesthetic infiltration of the palate during cleft palate repair is universally practiced. The benefits of local anesthetic infiltration are twofold: to provide anesthesia to the terminal branches of the nasopalatine and greater palatine nerves that are in the immediate area of the injection sites and to achieve hemostasis during closure when the medication is mixed with epinephrine. To administer local anesthetic infiltration of the palate, a 25 gauge needle is inserted next to the incision into the soft tissue. The tissue is first aspirated to determine safety of injection at that site. The medication is then injected parallel to the incision on both sides.
  Arms: Local anesthetic infiltration of the palate

SUMMARY:
Increased pain after cleft palate surgery is the leading cause of increased hospital length of stay, delayed oral intake, readmission, and respiratory compromise. The goal is to improve all outcomes by identifying the most effective evidenced-based method of intra-operative pain control.

DETAILED DESCRIPTION:
Cleft palate repair is associated with significant perioperative pain that may require increased depth of anesthesia intraoperatively and can interfere with oral intake and accentuate breathing difficulties postoperatively, resulting in increased length of hospital stay. Optimizing pain control in the perioperative period is essential to best practice for cleft palate repair. Infiltration of the palate with local anesthetic has long been the established mechanism for pain control to minimize intraoperative anesthetic requirement and postoperative opioid use. Suprazygomatic maxillary nerve block (SMB) administered immediately prior to cleft palate repair by anesthesiologists with fellowship training in regional anesthesia is an emerging technique for local anesthetic infiltration. The latter technique is thought to provide superior pain control due to its precise and targeted action on the nerves that innervate the palate, and because it is felt that duration of action may also be prolonged due to specific infiltration around these nerves as opposed to generalized infiltration in the palatal soft tissues. The goal of our study is to evaluate outcomes following the two routes for anesthetic infiltration during cleft palate repair. If either technique is found to be more effective or of greater duration, this can have direct impact in decreasing the need for perioperative opioid use, decreasing hospital length of stay, and less potential for airway suppression from excessive use of postoperative analgesics.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary cleft palate repair at Ann & Robert H. Lurie Children's Hospital of Chicago during the enrollment period. The typical child at the time of cleft palate repair is age 11 to 12 months.

Exclusion Criteria:

* Children with a known allergy to local anesthesia (i.e., ropivacaine or bupivacaine).
* Children with prior surgical repair of the palate.

Ages: 9 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of ultrasound-guided bilateral suprazygomatic maxillary nerve block on postoperative pain scores. | 48 hours after discharge
  The primary outcome for this aim will be pain scores, as determined by the Face, Legs, Activity, Crying, and Consolability scale. Minimum value is 0, maximum value is 10. Higher scores indicate more pain and therefore a worse outcome.
Evaluation of ultrasound-guided bilateral suprazygomatic maxillary nerve block on perioperative analgesia requirements. | 48 hours after discharge
  The primary outcome for this aim will be perioperative opioid consumption reported in morphine milligram equivalents.

SECONDARY OUTCOMES:
Evaluation of ultrasound-guided bilateral suprazygomatic maxillary nerve block on length of stay. | 48 hours after discharge
  A blinded researcher will perform a thorough review of patient data to determine the duration of hospital stay (hours).
Evaluation of ultrasound-guided bilateral suprazygomatic maxillary nerve block on time to oral intake. | 48 hours after discharge
  A blinded researcher will perform a thorough review of patient data to determine the time to oral intake (minutes).
Evaluation of ultrasound-guided bilateral suprazygomatic maxillary nerve block on total amount of fluids consumed. | 48 hours after discharge
  A blinded researcher will perform a thorough review of patient data to determine the total amount of fluids consumed (ounces).

CONTACTS AND LOCATIONS:
Overall Officials: Arun K Gosain, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No